CLINICAL TRIAL: NCT03729635
Title: Ultrasound-guided Pectoral-intercostal Fascial Plane Block for Patients With Severe Pain After Coronary Artery Bypass Graft Surgery: A Feasibility Study
Brief Title: Pectoral-Intercostal Fascial Plane Block Study
Acronym: PIFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Prabhakar, Clinical Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H17-03322
Record Dates: First submitted 2018-05-01; First posted 2018-11-05 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia, Regional; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PIFB performed to treat PSP (Experimental): Pectoral-intercostal fascial plane block (PIFB) is performed on patients with severe post-sternotomy pain (PSP) after coronary artery bypass graft surgery (CABG).
  Interventions: Procedure: Pectoral-intercostal fascial plane block (PIFB)

INTERVENTIONS:
Procedure: Pectoral-intercostal fascial plane block (PIFB) — Local anesthetic is infiltrated into the fascial plane between pectoralis major and the intercostal muscles lateral to the sternum to anesthetize the anterior cutaneous branches of the intercostal nerves.

SUMMARY:
Pain along the sternum following opening of the chest cavity, also known as post-sternotomy pain (PSP), is a common complication after heart surgery that is associated with several negative side effects. Unfortunately, an effective and safe treatment has not yet been discovered for PSP. However, recently a regional anesthesia technique called the pecto-intercostal fascial block (PIFB) was found to be associated with improved pain relief for breast surgery. The investigators plan to assess the feasibility of using PIFB as an effective and safe treatment for PSP.

DETAILED DESCRIPTION:
Post-sternotomy pain (PSP) is a common complication after cardiac surgery, occurring up to 49% of patients at rest according to one prospective study. In addition to decreased patient satisfaction, PSP has been associated with adverse post-operative events including delirium, hypertension, tachycardia, arrhythmias, respiratory complications and persistent post-surgical pain.

While most PSP can be effectively managed with opioids, non-steroidal anti-inflammatory drugs (NSAIDs) or central neuraxial blockades, these analgesia techniques also carry a high incidence of adverse effects. The use of opioid analgesics, for example, can contribute to respiratory depression, nausea, and delirium. While NSAIDs can be effective analgesics, they are also associated with postoperative kidney injury after cardiac surgery, a significant risk factor for mortality. Further, intrathecal or epidural techniques have a significant failure rate, and may be associated with severe hypotension, and devastating consequences such as neuraxial hematoma or infection. As such, alternative methods that are effective and safe for treating severe PSP remain elusive.

Peripheral regional anesthetic techniques have been demonstrated to reduce opioid consumption and may also provide improved respiratory mechanics. The pecto-intercostal fascial block (PIFB) was recently described in a descriptive letter by de la Torre and colleagues for anesthesia during breast surgery. In this technique, local anesthetic is infiltrated into the fascial plane between pectoralis major and the intercostal muscles lateral to the sternum to anesthetize the anterior cutaneous branches of the intercostal nerves. While the authors do state improved analgesia for breast surgery in their experience with use of this block, specific outcomes such as pain scores or opioid consumption are not reported.

The anterior cutaneous branches of the T2 to T6 intercostal nerves are thought to be the major sensory innervators of the sternum.

Using the same PIFB described above, the investigators have recently treated a patient successfully with severe PSP after CABG. To our knowledge, there is limited literature describing the use of this block for treatment of PSP. The investigators plan to conduct a prospective feasibility study to 1) assess the feasibility of using PIFB to reduce PSP in post-coronary bypass and/or valvular surgery patients and 2) obtain subjective data with regard to patient satisfaction and reduction in opioid consumption use that may help guide future, well-powered, randomized studies. 3) Describe any adverse outcomes following PIFB.

The study will be a prospective observational cohort study of twenty patients who are undergoing sternotomy for coronary bypass and/or valvular surgery. This is a proof-of-concept study with no prospective literature with respect to PIFB use in PSP post-cardiac surgery to guide sample size estimation. A minimum sample size of 12 patients has been recommended for pilot studies. By convenience sampling, the investigators have chosen to study 20 patients to demonstrate feasibility.

On the day of surgery, patients admitted to St. Paul's Hospital for cardiac procedure will be checked-in by a surgical nursing staff prior to the operation. During this time, the nursing staff will ask if the patient would like to learn more about the study and whether the patient is comfortable being approached by a member of the study group. If the patient agrees, a study team member will approach the patient and explain what the study entails, why the investigators are doing the study and how it may affect his/her care. The investigators will seek verbal permission to re-approach for recruitment following the surgery if the pain is moderate to severe. Those who are interested and gives verbal permission to be reapproached would be noted in the chart.

After the surgery, nursing staff in the Cardiac Surgery Intensive Care Unit (CSICU) who are looking after patients who have been extubated, are oriented (Confusion Assessment Method [CAM] negative and Richmond Agitation Scale [RASS] of +1 to -2), and are complaining of moderate to severe pain (>5/10 NPRS) related to the sternal area will contact a study team member. After verifying that the patient has given permission to be reapproached, a study team member will reconfirm interest in participating in the study and obtain a written consent prior to commencing the block. Subjects will be clearly informed that they will be free to discontinue participation in the study at any time. The investigators are responsible for ensuring that signed informed consent is obtained from all patients before enrolment.

After written informed consent, subjects will officially be de-identified by means of having a subject number assigned to them by which they will henceforth be identified in the study.

The principal investigator will assure that appropriate training relevant to the study is given to the medical, nursing, and other staff involved. The PIFB will be performed only by experienced regional anesthesiologists that have performed more than 200 ultrasound-guided peripheral nerve blocks.

Intravenous access, invasive blood pressure measurements, continuous electrocardiography and oxygen saturation monitoring will be confirmed throughout the procedure and for at least 60 minutes afterwards. Pre-block NPRS and opioid consumption over the hours between surgery and block will be recorded. Light sedation as required/indicated will be provided as per routine clinical practice with boluses of midazolam (0.01-0.03 mg/kg) and fentanyl (0.25-1.0 mcg/kg), with the goal of maintaining verbal contact with the patient throughout the procedure.

A GE LOGIQ e ultrasound machine (GE Healthcare Technologies, Waukesha, Wisconsin, USA) and a 12 Megahertz (MHz) ultrasound probe will be used for all blocks in the study. The probe will be prepared with a sterile probe covering. The patient's skin will be prepared with a 2% chlorhexidine antiseptic solution.

PIFB Procedure:

PIFB will be performed as described in the literature. The patient will be positioned supine. Using ultrasound guidance, a parasagittal view approximately 2.5cm lateral to the sternum will be obtained. After optimal imaging of pectoralis major muscles (PMM), the ribs/sterno-costal cartilage, and internal intercostal muscle (IIM) has been obtained, a 25 gauge hypodermic needle will be used to infiltrate the skin and subcutaneous tissues with 1% lidocaine, starting caudad to the ultrasound probe in a direction cephalad into the PMM. Using an in-plane technique, a 80-100 mm 22 gauge insulated regional block needle (Pajunk) will be inserted through the skin inferior to the probe and directed cephalad toward the fascial plane deep to PMM and superficial to the IIM and ribs/sterno-costal cartilage. The needle will be guided under ultrasound visualization towards the above-described plane. Local anesthetic will be injected initially at this location ensuring interfascial spread and not intramuscular injection. The needle will be redirected cephalad to ensure local is administered into the plane at each interspace from approximately T5-T6 cephalad to T2-T3. If required the needle will be removed and re-inserted at a cephalad position. A total of 20 ml of 0.25% ropivacaine will be injected in increments, using frequent aspiration to test for inadvertent intravascular needle placement. The PIFB will then be repeated on the contralateral side. A maximum total of 40 ml of 0.25% ropivacaine will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a CABG and/or valve Surgery.
* Extubated and on no assisted ventilation
* NPRS equal to or greater than 5 related to sternal pain despite standard treatment
* Aged 19-80
* American Society of Anesthesiologists Physical Status Classification System 1 to 4 (ASA I-IV)
* Provided written informed consent
* Body Mass Index < 35 kg/m^2
* Patient weight equal to or greater than 50 kg
* CAM negative and RASS of +1 (restless) to -2 (light sedation)

Exclusion Criteria:

* A known history or allergy, sensitivity, or any other form of reaction to amide-type local anesthetics.
* Suspected inability to comply with study procedures, including language difficulties, or medical history and/or concomitant disease, as judged by the investigator.
* A neurological and/or vascular condition which may preclude eligibility for peripheral nerve blockade as judged by the investigator.
* Coagulopathy
* Previous inclusion in this study.
* Participation in other clinical studies during this study or in the 14 days prior to admission to this study.
* Neuromuscular disease
* Thoracotomy
* Mini-Sternotomy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of PIFB in reduction of PSP following Sternotomy | Baseline to 30 minutes post-block completion
  Defined as successful reduction of NPRS by 2 or more points

SECONDARY OUTCOMES:
Numeric pain rating score (NPRS) | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  One NPRS related to post-sternotomy pain and one NPRS related to other pain (0-10 scale range, 0=no pain, 10=worst possible pain)
Opioid and analgesic use | 24 hours after block or until discharge from Cardiac Surgery Intensive Care Unit (CSICU) (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Dose of opioid and analgesics used before and after block
Duration of block | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Defined as time to first rescue analgesic
Blood pressure | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Patient blood pressure (systolic and diastolic) as shown on the vital signs monitor
Vasopressor medications administered | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Type of vasopressors given after the block (if any)
Dose of Vasopressor medications administered | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Dose of vasopressors given after the block (if any)
Heart rate | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Patient heart rate as shown on the vital signs monitor
Respiration Rate (RR) | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Patient RR as shown on the vital signs monitor
Peripheral Capillary Oxygen (SPO2) | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Patient SpO2 as shown on the vital signs monitor
Supplemental Oxygen (O2) | Baseline to 24 hours after block or until discharge from CSICU (data collection times: at 5, 10, 20, 30 minutes, 1 hour, 2 hours and every 2 hours after that from time of block)
  Patient O2 as shown on the vital signs monitor (if any)
Most Painful Site | 30 minutes 12 hours and 24 hours post block if still in CSICU
  Patients are asked to identify the area where they feel the most pain. No scale is used, just verbal indication or by pointing to the area.
Confusion Assessment Method (CAM) | 12 hours and 24 hours post block (if still in CSICU)
  A valid method of monitoring/diagnosing delirium in intensive care unit patients The diagnosis of delirium by CAM requires the presence of three of the four features listed (A: Acute onset and Fluctuating course; B: Inattention; C: Disorganized thinking; D: Altered level of consciousness)
Loss of Sensation | 30 minutes post block
  The Anesthesiologist will assess if there is a loss of sensation along the sternotomy. This is done by asking if the patient can feel cold in different areas of the chest. There is no scale for this measure, it is recorded as yes or no with a description if the assessor feels it is necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD, Study Chair — University of British Columbia; Kevin Rondi, MD, Study Chair — University of British Columbia; Simon Bruce, MD, Study Chair — University of British Columbia; James Abel, MD, Study Chair — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Background] Huang AP, Sakata RK. Pain after sternotomy - review. Braz J Anesthesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjane.2014.09.013. Epub 2016 Apr 23. PMID 27343790
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825
- [Background] Brown JR, Cochran RP, MacKenzie TA, Furnary AP, Kunzelman KS, Ross CS, Langner CW, Charlesworth DC, Leavitt BJ, Dacey LJ, Helm RE, Braxton JH, Clough RA, Dunton RF, O'Connor GT; Northern New England Cardiovascular Disease Study Group. Long-term survival after cardiac surgery is predicted by estimated glomerular filtration rate. Ann Thorac Surg. 2008 Jul;86(1):4-11. doi: 10.1016/j.athoracsur.2008.03.006. PMID 18573389
- [Background] Barr AM, Tutungi E, Almeida AA. Parasternal intercostal block with ropivacaine for pain management after cardiac surgery: a double-blind, randomized, controlled trial. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):547-53. doi: 10.1053/j.jvca.2006.09.003. Epub 2006 Dec 22. PMID 17678782
- [Background] McDonald SB, Jacobsohn E, Kopacz DJ, Desphande S, Helman JD, Salinas F, Hall RA. Parasternal block and local anesthetic infiltration with levobupivacaine after cardiac surgery with desflurane: the effect on postoperative pain, pulmonary function, and tracheal extubation times. Anesth Analg. 2005 Jan;100(1):25-32. doi: 10.1213/01.ANE.0000139652.84897.BD. PMID 15616047
- [Background] de la Torre PA, Garcia PD, Alvarez SL, Miguel FJ, Perez MF. A novel ultrasound-guided block: a promising alternative for breast analgesia. Aesthet Surg J. 2014 Jan 1;34(1):198-200. doi: 10.1177/1090820X13515902. No abstract available. PMID 24396082
- [Background] Warner L, Ritter MJ. 2017. Bilateral Pecto-Intercostal Fascial Plane Block for Acute Relief of Post-Sternotomy Pain. Scientific Abstracts and ePosters: ASRA 42nd Annual Regional Anesthesiology and Acute Pain Medicine Meeting April 6-8, 2017 San Francisco, CA. Reg Anesth Pain Med. 2017; 42 (6): 802-818.
- [Background] Liu V, Mariano ER, Prabhakar C. Pecto-intercostal Fascial Block for Acute Poststernotomy Pain: A Case Report. A A Pract. 2018 Jun 15;10(12):319-322. doi: 10.1213/XAA.0000000000000697. PMID 29293481
- [Background] Scientific Abstracts and ePosters: ASRA 42nd Annual Regional Anesthesiology and Acute Pain Medicine Meeting April 6-8, 2017 San Francisco, CA. Reg Anesth Pain Med. 2017; 42 (6): 802-818.
- [Background] Del Buono R, Costa F, Agro FE. Parasternal, Pecto-intercostal, Pecs, and Transverse Thoracic Muscle Plane Blocks: A Rose by Any Other Name Would Smell as Sweet. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):791-792. doi: 10.1097/AAP.0000000000000464. No abstract available. PMID 27776103
- [Background] Julious, SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceut Statist. 2005;4:287-291.
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804